CLINICAL TRIAL: NCT00521339
Title: A Phase 2, Open-label Multi-center Study to Evaluate the Safety, Pharmacodynamics, Pharmacokinetics, and Efficacy of Apremilast in Subjects With Recalcitrant Plaque-type Psoriasis
Brief Title: Apremilast Safety and PK Study in Recalcitrant Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-004
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis-Type Psoriasis; Plaque-Type Psoriasis
Keywords: Apremilast,; Psoriasis,; PASI-75,; sPGA
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apremilast 20 mg BID/ 30 mg BID (Experimental): Apremilast 20 mg or 30 mg orally twice per day
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — 20 mg PO (by mouth) twice per day (BID) for 84 days and then an additional 84 days during the optional treatment extension period. For subjects meeting the dose escalation criteria, dosage during the optional treatment extension period can be increased to 30 mg BID.
  Other Names: Otezla; CC-10004

SUMMARY:
The study will test the safety and tolerability of Apremilast twice a day in participants with recalcitrant plaque type psoriasis.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, open-label, study to evaluate the safety, tolerability, pharmacodynamics, pharmacokinetics and efficacy of Apremilast in participants with recalcitrant plaque-type psoriasis.

Approximately 31 participants were enrolled and received 20 mg apremilast orally BID and, in participants who are non-responders after 84 days of apremilast, 30 mg Apremilast over the course of the two study treatment phases. The study consisted of four phases: Screening Phase - up to 35 days, Treatment Phase of 84 days, Extension Phase of 84 days and a Observational Follow-up Phase of 28 days.

During the Treatment Phase, participants received two 20 mg Apremilast capsules each day. Following the Treatment Phase, participants had the option to continue on treatment during the Extension Phase. During the Extension Phase, participants either continued to take two 20 mg or dose escalated to two 30 mg of Apremilast each day. Participants who were considered responders (achieved a Psoriasis Area and Severity Index (PASI-75) at the beginning of the Extension Phase continued on 20 mg twice per day (BID) while the remaining participants received 30 mg capsules BID. The Extension Phase was introduced after some participants had already completed the study; therefore, there were several participants who never had the opportunity to continue into the Extension Phase. All participants were asked to participate in a 4-week post-treatment observational follow-up phase either upon completion of the study or upon discontinuation of study drug for those participants who terminated the study early.

ELIGIBILITY:
Inclusion Criteria:

Must understand and voluntarily sign an informed consent form

* Must be male or female subject of any ethnic origin or race that is >18 years at time of consent
* Must have a documented history of plaque-type psoriasis for at least 6 months prior to screening visit
* Subjects must fulfill criteria outlined in at least one of the following clinical categories:

  * Unresponsive to standard systemic therapy, as defined by clinical history, in the investigator's opinion, i.e. inadequate response to one or more adequate treatment course (s) of standard systemic therapy
  * Intolerant to or cannot receive (e.g., contraindication to prescribe) standard systemic therapy or biological interventions for psoriasis
* Must have a Static Physician Global Assessment (sPGA) score of at least 3 and a Body surface area (BSA) ≥ 10% at screening
* Must meet the specified laboratory criteria:

  o Must be able to adhere to the study visit schedule and study protocol requirements
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening (Visit 1). In addition, FCBP must agree to use two of the following adequate forms of contraception methods such as oral, injectable, or implantable hormonal contraception; tubal ligation; intrauterine device; barrier contraceptive with spermicide or vasectomized partner while on study. A FCBP must agree to have pregnancy tests every 4 weeks while on study medication.
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with FCBP

Exclusion Criteria:

* History of clinically significant (as determined by the investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major disease
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or lactating females
* History of active tuberculosis (TB) infection within 3 years prior to the screening visit. Infections which occurred > 3 years prior to entry must have been effectively treated
* History of incompletely treated latent (as indicated by a positive PPD [purified protein derivative] skin results) TB infection
* Clinically significant abnormality on the chest x-ray (CXR) at screening
* Psoriasis flare within 30 days of screening, as defined by protocol
* Use of systemic therapy for psoriasis within 28 days of Visit 2 (Baseline).
* Topical therapy as defined in the protocol Adalimumab, etanercept, efalizumab or infliximab use within 56 days of Visit 2 (Baseline)
* Alefacept use within 180 days of Visit 2 (Baseline)
* Phototherapy Ultraviolet light A (UVA), Ultraviolet light B (UVB), Psoralens and long-wave ultraviolet radiation (PUVA) within 28 days of Visit 2 (Baseline)
* Use of any investigational drug within 28 days of Visit 2 (Baseline), or 5 half lives if known (whichever is longer) Clinically significant abnormality on 12-lead Electrocardiogram (ECG) at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - Tufts-New England Medical Center Hospitals, Boston, Massachusetts
  - Central Dermatology, St Louis, Missouri
  - Oregon Medical Research Center, P.C., Portland, Oregon
  - Baylor Research Institute, Dallas, Texas

REFERENCES:
- [Result] Gottlieb AB, Matheson RT, Menter A, Leonardi CL, Day RM, Hu C, Schafer PH, Krueger JG. Efficacy, tolerability, and pharmacodynamics of apremilast in recalcitrant plaque psoriasis: a phase II open-label study. J Drugs Dermatol. 2013 Aug;12(8):888-97. PMID 23986162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants must have had a diagnosis of plaque-type psoriasis for at least 6 months and had an insufficient response, were unresponsive, intolerant of, or had medical contraindications to standard systemic therapy or biological treatment for plaque-type psoriasis. The study was conducted at 4 sites in the U.S. from 20 August 2007 to 12 May 2009.
Pre-assignment Details: The study consisted of a 12-week treatment phase, a 12-week treatment extension phase and a 4-week observational follow-up phase. Participants could enter the follow-up phase at any time during the study. Some participants had completed the study before the extension phase was added and therefore never had the opportunity to participate.
Groups:
- Apremilast 20mg: Participants received 20mg Apremilast capsules by mouth (PO) twice a day (BID) on Days 1 through 85 during the Treatment Phase
- Apremilast 20mg/20mg: Participants who received 20 mg apremilast BID during the treatment phase (Weeks 0-12) who were responders (achieved a 75% reduction in the Psoriasis Area Severity Index [PASI-75]) continued to receive 20 mg apremilast BID during the 12-week extension phase (Weeks 12-24).
- Apremilast 20mg/30mg: Participants who received 20 mg apremilast BID during the treatment phase (Weeks 0-12) who were non-responders (did not achieve PASI-75 response) received 30 mg apremilast BID during the 12-week extension phase
Period: Treatment Phase
Arm/Group | Apremilast 20mg | Apremilast 20mg/20mg | Apremilast 20mg/30mg
Started | 31 | 0 | 0
Received Apremilast | 30 (1 participant withdrew consent prior to first visit and was excluded from safety population) | 0 | 0
Completed | 19 | 0 | 0
Not Completed | 12 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Intolerability to study drug | 2 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Treatment Extension Phase
Arm/Group | Apremilast 20mg | Apremilast 20mg/20mg | Apremilast 20mg/30mg
Started | 0 | 4 (Some participants had completed the treatment phase prior to inception of extension phase) | 7 (Some participants had completed the treatment phase prior to inception of extension phase)
Completed | 0 | 4 | 4
Not Completed | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Death | 0 | 0 | 1
Period: Observational Follow Up Phase
Arm/Group | Apremilast 20mg | Apremilast 20mg/20mg | Apremilast 20mg/30mg
Started | 14 | 4 | 4
Completed | 14 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who were enrolled and received at least one dose of study medication.
Groups:
- Apremilast 20 mg (Treatment Phase): Apremilast 20mg capsules by PO BID for Days 1 through 85 administered during the treatment phase
Arm/Group | Apremilast 20 mg (Treatment Phase)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Recalcitrant Psoriasis History [Mean (Standard Deviation); unit: years] — Eligible participants had a diagnosis of plaque-type psoriasis at least 6 months prior to screening and either had an insufficient response, were unresponsive to, were intolerant of, or had medical contraindications to standard systemic therapy or biological treatment for plaque-type psoriasis. Participants also had a Static Physician Global Assessment (sPGA) score of at least 3 and psoriasis affected body surface area (BSA) involvement ≥ 10% at screening. The sPGA is a measure of psoriasis disease severity at the time of evaluation by the investigator.
  years | 10.9 (11.36)
Mean Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: units on a scale] — PASI: Combined assessment of lesion severity and area affected into single score; range: 0(no disease) to 72(maximal disease).
  units on a scale | 17.0 (6.77)
Mean Body Surface Area (BSA) Involvement [Mean (Standard Deviation); unit: Percentage of BSA] — The BSA estimate was based on the palm area of the hand of the participant which equates to 1% of the total body surface area.
  Percentage of BSA | 22.4 (13.85)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events (TEAEs) During the Treatment Phase
Description: TEAE = any AE occurring or worsening on or after the first treatment with any study drug. Related = suspected by investigator to be related to study treatment. National Cancer Institute [NCI] Common Toxicity Criteria for Adverse Events [CTCAE], Version 3.0, grades: 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, 5 = death.
  Adverse event (AE) = any noxious, unintended, or untoward medical occurrence occurring at any dose that may appear or worsen in a participant during the course of a study, including new intercurrent illness, worsening concomitant illness, injury, or any concomitant impairment of participant's health, including laboratory test values, regardless of etiology. Serious adverse event (SAE) = any AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect; constitutes an important medical event.
Time Frame: Week 0 to Week 12
Population: Safety population consisted of all participants who were enrolled and received at least one dose of study medication.
Measure: Number; unit: participants
Groups:
- Apremilast 20 mg: Apremilast 20mg capsules PO BID on Days 1 through 85 administered during the Treatment Phase
Arm/Group | Apremilast 20 mg
Number analyzed (Participants) | 30
participants
  ≥ 1 AE | 25
  ≥ 1 AE with a suspected relationship to study drug | 13
  ≥ 1 severe AE | 3
  ≥ 1Severe AE suspected to be related to study drug | 1
  ≥ 1 SAE | 0
  ≥ AE leading to study drug discontinuation | 4
  >=1 treatment-related AE drug discontinued | 2

2. Secondary Outcome: Percentage of Participants With at Least a 1 Point Reduction on 0 to 5 Point Scale From Baseline in Static Physician Global Assessment (sPGA) at Week 12
Description: The static Physician's Global Assessment (sPGA) rated the investigator's overall clinical assessment of a participants plaque thickness, erythema, and scaling on a 6-point scale ranging from 0 (clear, except for residual discoloration) to 5 (majority of plaques have severe thickness, erythema, and scale). To assign a sPGA score, the investigator examined all psoriatic lesions and assigned a severity score ranging from 0 to 5 for thickness, erythema, and scaling. Scores for thickness, erythema, and scaling are summed and the mean of these 3 scores equals the overall sPGA score. Decreases in sPGA correspond to clinical improvement.
Time Frame: Baseline and Week 12
Population: Safety population consisted of all participants who were enrolled and received at least one dose of study medication. Last Observation Carried Forward.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apremilast 20 mg PO BID (Treatment Phase): Apremilast 20mg capsules by mouth (PO) twice a day (BID) for Days 1 through 85 administered during the treatment phase
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 30
percentage of participants | 66.7 [47.2 to 82.7]

3. Secondary Outcome: Percent Change From Baseline in Psoriasis Area Severity Index (PASI) Score at Week 12
Description: The PASI score was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) was multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score.
Time Frame: Baseline and Week 12
Population: Safety population consisted of all participants who were enrolled and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Apremilast 20 mg: Apremilast 20mg capsules PO BID for Days 1 through 85 administered during the treatment phase
Arm/Group | Apremilast 20 mg
Number analyzed (Participants) | 20
percent change | -59.0 (31.59)

4. Secondary Outcome: Percentage of Participants Who Achieved a PASI-75 Score at Week 12
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 12. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the4 anatomic regions was scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) was multiplied by the degree of involvement for each anatomic region and then multiplied by a constant.
Time Frame: Baseline to Week 12
Population: Safety population consisted of all participants who were enrolled and received at least one dose of study medication. If participant had a missing evaluation for any time point assessments, the last observation carried forward (LOCF) method of imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 20 mg
Number analyzed (Participants) | 30
percentage of participants | 30.00 [14.7 to 49.4]

5. Secondary Outcome: Percentage of Participants Who Achieved a PASI-50 Score at Week 12
Description: PASI -50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score at Week 12. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head,trunk, upper limbs, and lower limbs. Degree of involvement on each of the4 anatomic regions was scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) was multiplied by the degree of involvement for each anatomic region and then multiplied by a constant.
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast 20 mg
Number analyzed (Participants) | 30
percentage of participants | 46.7 [28.3 to 65.7]

6. Secondary Outcome: Maximal PASI Response Documented for Each Participant During Treatment Phase
Description: PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head,trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score.
Time Frame: Baseline to Week 12
Population: Maximal PASI response was not analyzed since similar information was captured in change in psoriasis area severity Index (PASI) score at Day 85, which is week 12.
Groups:
- Apremilast 20 mg PO BID (Treatment Phase): Apremilast 20mg capsules by mouth (PO) twice a day (BID) am and pm for Days 1 through 85 administered during the Treatment Phase
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 0

7. Secondary Outcome: Percent Change From Baseline in the Psoriasis Affected Body Surface Area (BSA) Involvement at Week 12
Description: The BSA estimate was based on the palm area of the hand of the participant which equates to 1% of the total body surface area.
Time Frame: Baseline to Week 12
Population: Safety population consisted of all participants who were enrolled and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Percent change in BSA
Arm/Group | Apremilast 20 mg
Number analyzed (Participants) | 20
Percent change in BSA | -53.0 (35.50)

8. Secondary Outcome: Time to Clinically Relevant Response (Time to Achieve PASI-50) During Treatment Phase
Description: Time to clinically relevant response (time to achieve PASI-50) during treatment phase was not analyzed. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head,trunk, upper limbs, and lower limbs. Degree of involvement on each of the4 anatomic regions was scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) was multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score.
Population: Time to achieve PASI-50 was not analyzed since the study enrolled a small number of participants and the number of participants who achieved PASI-50 was even smaller.
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 0

9. Secondary Outcome: Time to Achieve PASI-75 During Treatment Phase
Description: Time to achieve PASI-75 during treatment phase was not analyzed. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the4 anatomic regions was scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) was multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score.
Population: Time to achieve PASI-75 was not analyzed, due to the small number of participants enrolled and who achieved PASI-75.
Groups:
- Apremilast 20 mg: Apremilast 20mg capsules by mouth (PO) twice a day (BID) for Days 1 through 85 administered during the treatment phase
Arm/Group | Apremilast 20 mg
Number analyzed (Participants) | 0

10. Secondary Outcome: Time to Relapse of Psoriasis (50% Loss of Maximal PASI Score Improvement in Participants Who Achieved at Least PASI-50 During the Treatment Phase) During the Observational Follow up Phase
Description: Time to relapse of psoriasis (50% loss of maximal PASI score improvement in participants who achieved at least PASI-50 during the treatment phase) during the observational follow up phase was not analyzed. Time to relapse of psoriasis was defined as a 50% loss of maximal PASI score improvement in participants who achieved at least PASI-50 during the treatment or extension phase. The lesion on each area of the body was assessed for redness, thickness, and scaling.
Time Frame: 28-day Observational Follow-up Phase; Days 168 to Day 196.
Population: Time to relapse of psoriasis was not analyzed due to the small number of participants enrolled and who achieved PASI-50 and entered the observation follow-up phase.
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 0

11. Secondary Outcome: Percent of Participants With Psoriatic Arthritis Who Achieved an American College of Rheumatology 20% Improvement (ACR-20) Response at Week 12
Description: A participant was a responder if the following 3 criteria for improvement from baseline were met:
  * ≥ 20% improvement in 78 tender joint count;
  * ≥ 20% improvement in 76 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters: Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Patient's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); C-Reactive Protein.
Time Frame: Baseline to Week 12
Population: Safety population consisted of all participants who were enrolled and received at least one dose of study medication. Last observation carried forward was used. Only a small percentage of participants had psoriatic arthritis.
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 8
percentage of participants | 25.0

12. Secondary Outcome: Time to Relapse of Psoriatic Arthritis During the Observational Follow-up Phase
Description: A relapse was defined as a 50% loss of maximal American College of Rheumatoid (ACR) Score improvement in participants with psoriatic arthritis who achieved at least an ACR 20 score during the treatment phase.
  Relapses were only captured prior to the prescription of concomitant psoriatic treatment.
Time Frame: Observational follow up phase; Days 168 to Day 196
Population: This endpoint was not summarized since there were only 8 participants with psoriatic arthritis enrolled in the study and only 2 participants who achieved an ACR 20 response during the treatment phase.
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 0

13. Secondary Outcome: Area Under the Plasma Concentration Time-curve From 0 to 12 Hours Post Dose (AUC 0-12)
Description: Plasma concentrations of apremilast were determined using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). For Day 1, AUC0-12 was calculated, using linear trapezoidal area method in WinNonlin (linear-linear trapezoidal). For Days 85 and 169/170, the AUC during a dosing interval (12 hours) (AUC0-12), was calculated at steady-state using the partial area function within WinNonlin.
  .
Time Frame: Day 85 Pre-dose, 0.5, 1, 2, 4, 8, and 12 hours after the AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for Apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Apremilast 20mg: Apremilast 20mg capsules by PO BID for Days 1 through 85 administered during the treatment phase
Arm/Group | Apremilast 20mg
Number analyzed (Participants) | 10
ng*hr/mL | 2424.48 (46.87)

14. Secondary Outcome: Peak (Maximum) Plasma Concentration of Medication (Cmax)
Description: The maximum observed plasma concentration of apremilast (Cmax); the maximum plasma concentration (Cmax) was obtained directly from the observed concentration-time data on Days 1, 85, and 169/170, respectively.
Time Frame: Day 85 Pre-dose, 0.5, 1, 2, 4, 8, and 12 hours after the AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for Apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Apremilast 20mg
Number analyzed (Participants) | 10
ng/mL | 364.85 (38.25)

15. Secondary Outcome: Trough Plasma Concentration (Cmin)
Description: The trough observed plasma concentration of apremilast (Cmin) was determined directly from the observed pre-AM dose concentration on Day 85.
Time Frame: Day 85 Pre-dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Apremilast 20mg
Number analyzed (Participants) | 10
ng/mL | 101.36 (71.6)

16. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) During the Treatment Phase
Description: The time to reach Cmax (Tmax) was obtained directly from the observed concentration-time data on Day 85. Actual times utilized were used for reporting Tmax values.
Time Frame: Day 85 Pre-dose, 0.5, 1, 2, 4, 8, and 12 hours after the AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast.
Measure: Median (Full Range); unit: hours
Arm/Group | Apremilast 20mg
Number analyzed (Participants) | 10
hours | 2.00 [1.00 to 4.03]

17. Secondary Outcome: Terminal Phase Elimination Half Life of Apremilast (t½)
Description: Terminal phase elimination half-life (t1/2) was calculated as follows: t1/2 = 0.693/λz. The terminal elimination rate constant (λZ) was estimated by linear regression of the log-transformed concentration-time data.
Time Frame: Day 85 Pre-dose, 0.5, 1, 2, 4, 8, and 12 hours after the AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Apremilast 20mg
Number analyzed (Participants) | 3
Liters | 7.832 (26.031)

18. Secondary Outcome: Apparent Total Clearance of Apremilast From Plasma After Extravascular Administration (CLz/F) During the Treatment Phase
Description: The apparent total clearance of apremilast from plasma after extravascular administration (CLz/F); for Day 1, apparent clearance of drug from plasma (CL/F) was not calculated.
  For Day 85, Apparent clearance of drug from plasma after extravascular administration (CL/F) was calculated as follows: CL/F= Dose/AUC^12 where τ=12.
Time Frame: Day 85 Pre-dose, 0.5, 1, 2, 4, 8, and 12 hours after the AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast. This analysis was performed for participants with normal renal function only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hour
Arm/Group | Apremilast 20mg
Number analyzed (Participants) | 3
mL/hour | 8249.19 (46.87)

19. Secondary Outcome: Apparent Total Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F) During the Treatment Phase
Description: Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) (for Days 1, 85, and 169/170)
  1. For Day 1, Vz/F was not calculated.
  2. For Days 85 and 169/170, apparent volume of distribution of drug (V/z) based on the terminal phase was calculated as follows: Vz/F=Dose/(λ*AUC^12)
Time Frame: Day 85
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Apremilast 20mg
Number analyzed (Participants) | 3
mL | 107616.08 (47.03)

20. Secondary Outcome: Accumulation Index (R)
Description: Accumulation represents the relationship between the dosing interval and the rate of elimination for the drug.
Time Frame: Day 85 Pre-dose, 0.5, 1, 2, 4, 8, and 12 hours after the AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Apremilast 20mg
Number analyzed (Participants) | 10
ratio | 1.68 (53.17)

21. Secondary Outcome: Mean Residence Time (MRT) During the Treatment Phase
Description: Mean Residence Time (MRT) is defined as the mean duration of time the drug spends in the body. The average concentration at steady state (Cavg) (for Day 85 was calculated as follows: Cavg = (Day 85 AUC0-12)/(12).
Time Frame: Day 85 Pre-dose, 0.5, 1, 2, 4, 8, and 12 hours after the AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Apremilast 20mg PO BID: Apremilast 20mg capsules by PO BID for Days 1 through 85 administered during the treatment phase
Arm/Group | Apremilast 20mg PO BID
Number analyzed (Participants) | 10
hours | 202.04 (46.87)

22. Secondary Outcome: Change From Baseline in Peripheral Blood T Cell, B Cell, and NK Cell Subsets at Week 12
Description: T cells or T lymphocytes, a type of white blood cell, play a role in cell-mediated immunity. T cells are distinguished from other lymphocytes by the presence of a T-cell receptor (TCR) on the cell surface and mature in the thymus. B cells, a type of lymphocyte in the humoral immunity of the adaptive immune system can be distinguished by the presence of a protein on the B cells outer surface called a B cell receptor (BCR). This receptor protein allows a B cell to bind to a specific antigen and make antibodies against antigens [(antigen-presenting cells APCs)], and to develop into memory B cells after activation by antigen interaction. Natural Killer Cells (NK) are a type of cytotoxic lymphocyte critical to the innate immune system. Their role is analogous to that of cytotoxic T cells in the vertebrate adaptive immune response. They constitute the third kind of cells differentiated from the common lymphoid progenitor generating B and T lymphocytes and mature in the bone marrow.
Time Frame: Baseline and Week 12
Population: Population includes participants who took at least 1 dose of study medication and were measured for the peripheral blood T cell, B cell and NK cell subsets at Baseline and Week 12.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 30
percentage of lymphocytes
  CD 16 + CD 56 (NK cells) | -0.7 (3.05)
  CD 19 (B-cells) | -0.5 (2.63)
  CD 3 (T-cells) | 0.6 (2.63)

23. Secondary Outcome: Percent Change From Baseline of CD3 in the Dermis of the Psoriatic Skin Biopsy at Week 12
Description: The aim of the study was to measure the pharmacodynamic effects of apremilast in participants with plaque psoriasis in skin affected by psoriasis, immune cells enter the skin through blood vessels and cause the epidermis to grow very rapidly and to stop shedding properly. This causes thickening of the skin as well as the scaly build up composed of dead skin cells seen on areas affected by psoriasis.
Time Frame: Baseline and Week 12
Population: Population includes participants who took at least 1 dose of study medication and were measured for the Psoriatic Skin Biopsy at Baseline and Week 12. Participation was optional for the pharmacodynamic portion of the study.
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 16
percent change | -62.0 [-84.3 to 290.9]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Percent Change From Baseline of CD3 in the Epidermis of the Psoriatic Skin Biopsy at Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 16
percent change | -47.4 [-100.0 to 159.5]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.074, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Percent Change From Baseline of CD 11c in the Dermis of the Psoriatic Skin Biopsy at Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 15
percent change | -54.6 [-88.8 to 284]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.018, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Percent Change From Baseline of CD11c in the Epidermis of the Psoriatic Skin Biopsy at Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 14
percent change | -88.6 [-100.0 to 46.3]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Percent Change From Baseline of CD56 in the Dermis of the Psoriatic Skin Biopsy at Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 16
percent change | -12.5 [-68.9 to 57.1]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.632, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Percent Change From Baseline of CD56 in the Epidermis of the Psoriatic Skin Biopsy at Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 13
percent change | -73.3 [-100.0 to 311.1]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.242, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Percent Change From Baseline of Langerin in the Dermis of Psoriatic Skin Biopsy at Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 13
percent change | -57.9 [-100.0 to 178.3]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.329, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Percent Change From Baseline of Langerin in the Epidermis of the Psoriatic Skin Biopsy at Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 16
percent change | 17.1 [-78.7 to 300.0]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.130, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Percent Change From Baseline of Epidermal Thickness in the Psoriatic Skin Biopsy at Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 23
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 15
percent change | -34.3 [-65.4 to 42.2]

32. Secondary Outcome: Percent Change From Baseline in the Inducible Nitric Oxide (iNOS) Inflammatory Marker in Psoriatic Skin Biopsies
Description: Inflammatory markers associated with psoriasis (using skin biopsies) were used to detect acute inflammation and as markers of treatment response. The inflammatory markers were measured using Reverse transcriptase polymerase chain reaction (RT-PCR) and the messenger Ribonucleic acid (mRNA) is being measured.
Time Frame: Baseline and Week 12
Population: Population includes participants who took at least 1 dose of study medication and were measured for the Inflammatory Marker in Psoriatic Skin Biopsies at Baseline and Week 12. Participation was optional for the pharmacodynamic portion of the study.
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 12
percent change | -100.0 [-100.0 to 55.9]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: Percent Change From Baseline in the Interleukin (IL) IL-22 Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 6
percent change | -100.0 [-100.0 to -44.5]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.031, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: Percent Change From Baseline in the p40 Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 8
percent change | -86.7 [-100.0 to 51.7]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.039, Wilcoxon (Mann-Whitney)

35. Primary Outcome: Treatment Emergent Adverse Events (TEAEs) During the Extension Phase
Description: TEAE = any AE occurring or worsening on or after the first treatment with any study drug. Related = suspected by investigator to be related to study treatment. National Cancer Institute [NCI] Common Toxicity Criteria for Adverse Events [CTCAE], Version 3.0, grades: 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, 5 = death.
  Adverse event (AE) = any noxious, unintended, or untoward medical occurrence occurring at any dose that may appear or worsen in a participant during the course of a study, including new intercurrent illness, worsening concomitant illness, injury, or any concomitant impairment of participant's health, including laboratory test values, regardless of etiology. Serious adverse event (SAE) = any AE which: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event.
Time Frame: Week 12 to Week 24
Population: Safety population consisted of all participants who were enrolled and received at least one dose of study medication in treatment Extension Phase.
Measure: Number; unit: participants
Groups:
- Apremilast 20mg/20mg (Extension Phase): Participants who received 20 mg apremilast BID during the treatment phase (Weeks 0-12) who were responders (achieved a 75% reduction in the Psoriasis Area Severity Index [PASI-75]) continued to receive 20 mg apremilast BID during the 12-week extension phase (Weeks 12-24).
- Apremilast 20mg/30mg (Extension Phase): Participants who received 20 mg apremilast BID during the treatment phase (Weeks 0-12) who were non-responders (did not achieve PASI-75 response) received 30 mg apremilast BID during the 12-week extension
Arm/Group | Apremilast 20mg/20mg (Extension Phase) | Apremilast 20mg/30mg (Extension Phase)
Number analyzed (Participants) | 4 | 7
participants
  ≥ 1 AE | 4 | 5
  ≥ 1 AE with a suspected relationship to study drug | 0 | 2
  ≥ 1 severe AE | 1 | 1
  ≥ 1 SAE | 0 | 1

36. Secondary Outcome: Percent Change From Baseline in the Defensin Beta 4 (DEFB4) Inflammatory Marker in Psoriatic Skin Biopsies
Description: Inflammatory markers associated with psoriasis (using skin biopsies) were used to detect acute inflammation and as markers of treatment response. The inflammatory markers were measured using Reverse transcriptase polymerase chain reaction (RT-PCR) and the messenger Ribonucleic acid (mRNA) i being measured.
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 11
percent change | -82.3 [-100.0 to 14.5]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.014, Wilcoxon (Mann-Whitney)

37. Secondary Outcome: Percent Change From Baseline in the keratin16 (K16) Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 15
percent change | -78.6 [-99.9 to 217.7]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.015, Wilcoxon (Mann-Whitney)

38. Secondary Outcome: Percent Change From Baseline in the pluripotent19 (P19) Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 15
percent change | -68.3 [-100.0 to 326.6]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.018, Wilcoxon (Mann-Whitney)

39. Secondary Outcome: Percent Change From Baseline in the IL8 Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 15
percent change | -66.5 [-100.0 to 136.2]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.018, Wilcoxon (Mann-Whitney)

40. Secondary Outcome: Percent Change From Baseline in the MX1 (Gene That Encodes the Interferon-induced p78 Protein) Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 12
percent change | -52.6 [-97.0 to -1.3]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

41. Secondary Outcome: Percent Change From Baseline in the IL17A Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 11
percent change | -49.4 [-100.0 to 76.8]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.031, Wilcoxon (Mann-Whitney)

42. Secondary Outcome: Percent Change From Baseline in the Tumor Necrosing Factor (TNF) Alpha Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Week 0 to Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 14
percent change | -42.7 [-100.0 to 242.9]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.217, Wilcoxon (Mann-Whitney)

43. Secondary Outcome: Percent Change From Baseline in the Interferon (INF) Gamma Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 13
percent change | -37.6 [-100.0 to 250.3]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.539, Wilcoxon (Mann-Whitney)

44. Secondary Outcome: Percent Change From Baseline in the IL10 Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 15
percent change | -26.5 [-100.0 to 565.0]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.169, Wilcoxon (Mann-Whitney)

45. Secondary Outcome: Percent Change From Baseline in the Chemokine Ligand (CXCL9) Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 12
percent change | -36.4 [-97.1 to 1021.2]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.339, Wilcoxon (Mann-Whitney)

46. Secondary Outcome: Percent Change From Baseline in the IL2 Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 10
percent change | -25.0 [-100.0 to 875.7]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.898, Wilcoxon (Mann-Whitney)

47. Secondary Outcome: Percent Change From Baseline in the Dendritic Cell (CD83) Inflammatory Marker in Psoriatic Skin Biopsies
Description: as for outcome 32
Time Frame: Baseline and Week 12
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 12
percent change | 14.2 [-98.5 to 162.1]
Statistical Analysis 1: Comparison: Apremilast 20 mg PO BID (Treatment Phase); Test type: Superiority or Other; p = 0.622, Wilcoxon (Mann-Whitney)

48. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) at Week 12
Description: DLQI was the dermatology-specific quality of life (QOL) measure used for the psoriatic population. The DLQI was a validated, self-administered, 10-item questionnaire that measures the impact of skin disease on a participants QoL, based on recall over the past week. Domains include symptoms, feelings, daily activities, leisure, work, personal relationships, and treatment. Possible responses for each of the 10 items are: not at all, a little, a lot, and very much. Each question is rated on a scale of 0 to 3 with a total range of 0 to 30. Higher scores indicate greater impact of disease on QOL
Time Frame: Baseline to Week 12
Population: Only those with both a baseline and final/termination visit assessment were included in the analyses of change from baseline. Safety population consisted of all participants who were enrolled and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 20 mg PO BID (Treatment Phase)
Number analyzed (Participants) | 30
units on a scale | -4.7 (8.66)

49. Secondary Outcome: Change From Baseline in the Medical Outcome Study Short Form 36-item Health Survey (SF-36) Scores, Mental and Physical Components to Week 12
Description: The SF-36 was a self-administered instrument consisting of 8 multi-item scales that assess 8 health domains: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. A higher score post-baseline is indicative of improvement in the disease state. The summary physical health score included physical functioning, role-physical, bodily pain and general health. The summary mental health score included: vitality, social functioning, role-emotional and mental health. The resulting score for each subscale is then standardized, to obtain values ranging from 0 to 100, with higher values indicating a better QOL.
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Apremilast 20 mg: Apremilast 20mg capsules by PO BID for Days 1 through 85 administered during the treatment phase
Arm/Group | Apremilast 20 mg
Number analyzed (Participants) | 15
units on a scale
  Mental Component | 0.8 (7.45)
  Physical Component | 2.4 (7.64)

50. Secondary Outcome: Area Under the Plasma Concentration Time-curve From 0 to 12 Hours Post Dose (AUC 0-12) During the Extension Phase
Description: Plasma concentrations of apremilast were determined using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS).
Time Frame: Day 169 pre-dose, 0.5, 1, 2, 4, 8 12, 24 and 36 hours after AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Apremilast 20/30mg BID: Participants who received 20 mg apremilast BID during the treatment phase (Weeks 0-12) who were non-responders (did not achieve PASI-75 response) received 30 mg apremilast BID during the 12-week extension phase
Arm/Group | Apremilast 20/30mg BID
Number analyzed (Participants) | 3
ng*hr/mL | 2019.71 (63.62)

51. Secondary Outcome: Peak (Maximum) Plasma Concentration of Apremilast (Cmax) During the Extension Phase
Description: The maximum observed plasma concentration of CC-10004 (Cmax); the maximum plasma concentration (Cmax) was obtained directly from the observed concentration-time data on Days 169/170.
Time Frame: Day 169 pre-dose, 0.5, 1, 2, 4, 8 12, 24 and 36 hours after AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for Apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Apremilast 20mg/30mg PO BID (Treatment + Extension Phase): Participants who received 20 mg apremilast BID during the treatment phase (Weeks 0-12) who were non-responders (did not achieve PASI-75 response) received 30 mg apremilast BID during the 12-week extension phase
Arm/Group | Apremilast 20mg/30mg PO BID (Treatment + Extension Phase)
Number analyzed (Participants) | 3
ng/mL | 320.35 (47.64)

52. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) During the Extension Phase
Description: The time to reach Cmax (Tmax) was obtained directly from the observed concentration-time data on Day 169/170. Actual times utilized were used for reporting Tmax values.
Time Frame: Day 169 pre-dose, 0.5, 1, 2, 4, 8 12, 24 and 36 hours after AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for Apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Apremilast 20mg BID/30mg PO BID (Treatment + Extension Phase): Participants who received 20 mg apremilast BID during the treatment phase (Weeks 0-12) who were non-responders (did not achieve PASI-75 response) received 30 mg apremilast BID during the 12-week extension phase
Arm/Group | Apremilast 20mg BID/30mg PO BID (Treatment + Extension Phase)
Number analyzed (Participants) | 3
hours | 1.59 (42)

53. Secondary Outcome: Terminal Phase Elimination Half Life of Apremilast (t½) During the Extension Phase
Description: as for outcome 17
Time Frame: Day 169 pre-dose, 0.5, 1, 2, 4, 8 12, 24 and 36 hours after AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for Apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Apremilast 20mg/30mg PO BID (Treatment + Extension Phase)
Number analyzed (Participants) | 3
hours | 6.287 (22.879)

54. Secondary Outcome: Apparent Total Clearance of Apremilast From Plasma After Extravascular Administration (CL/F) During the Extension Phase
Description: For 169/170, apparent clearance of drug from plasma after extravascular administration (CL/F) was calculated as follows: CL/F= Dose/AUC12
Time Frame: Day 169 pre-dose, 0.5, 1, 2, 4, 8 12, 24 and 36 hours after AM dose
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hour
Arm/Group | Apremilast 20mg/30mg PO BID (Treatment + Extension Phase)
Number analyzed (Participants) | 3
mL/hour | 14853.59 (63.62)

55. Secondary Outcome: Apparent Total Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F) During the Extension Phase
Description: For Days 169/170, apparent volume of distribution of drug (V/z) based on the terminal phase was calculated as follows: Vz/F=Dose/(λ*AUC12) where λ = the terminal elimination rate constant
Time Frame: Day 169 pre-dose, 0.5, 1, 2, 4, 8 12, 24 and 36 hours after AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Groups:
- Apremilast 20mg BID/30mg PO BID (Treatment + Extension Phase): Participants who received 20 mg apremilast BID during the treatment phase (Weeks 0-12) who were non-responders (did not achieve PASI-75 response) received 30 mg apremilast BID during the 12-week extension
Arm/Group | Apremilast 20mg BID/30mg PO BID (Treatment + Extension Phase)
Number analyzed (Participants) | 3
mL | 134734.60 (63.70)

56. Secondary Outcome: Accumulation Index During the Extension Phase
Description: Accumulation represents the relationship between the dosing interval and the rate of elimination for the drug.
Time Frame: Day 169 pre-dose, 0.5, 1, 2, 4, 8 12, 24 and 36 hours after AM dose
Population: Not able to calculate the Accumulation Index at this time point; insufficient data collection for this calculation.
Groups:
- Apremilast 20mg/30mg PO BID (Treatment + Extension Phase): Participants who received 20 mg apremilast BID during the treatment phase (Weeks 0-12) who were non-responders (did not achieve PASI-75 response) received 30 mg apremilast BID during the 12-week extension
Arm/Group | Apremilast 20mg/30mg PO BID (Treatment + Extension Phase)
Number analyzed (Participants) | 0

57. Secondary Outcome: Mean Residence Time (MRT) During the Extension Phase
Description: Mean Residence Time (MRT) is defined as the mean duration of time the drug spends in the body. The average concentration at steady state (Cavg) (for Days169/170) was calculated as follows: Cavg = (Day 169/170)/(12)
Time Frame: Day 169 pre-dose, 0.5, 1, 2, 4, 8 12, 24 and 36 hours after AM dose
Population: Pharmacokinetic (PK) Population, consisting of all participants with evaluable plasma concentration data for apremilast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Apremilast 20mg/30mg PO BID (Treatment + Extension Phase)
Number analyzed (Participants) | 3
hours | 168.3092 (63.6203)

ADVERSE EVENTS:
Time Frame: Days 1 to Day 196 visit; Adverse Events (AE) were reported from the first day of study drug treatment through the 28 day observational follow up period. Maximum exposure to study medication was 171 days.
Groups:
- Apremilast 20 mg (Treatment Phase): Apremilast 20mg capsules by mouth (PO) twice a day (BID) for Days 1 through 85 administered during the treatment phase
Arm/Group | Apremilast 20 mg (Treatment Phase) | Apremilast 20mg/20mg (Extension Phase) | Apremilast 20mg/30mg (Extension Phase)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/4 | 1/7
Other Adverse Events (participants affected / at risk) | 25/30 | 4/4 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast 20 mg (Treatment Phase) (N=30) | Apremilast 20mg/20mg (Extension Phase) (N=4) | Apremilast 20mg/30mg (Extension Phase) (N=7)
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast 20 mg (Treatment Phase) (N=30) | Apremilast 20mg/20mg (Extension Phase) (N=4) | Apremilast 20mg/30mg (Extension Phase) (N=7)
NASOPHARYNGITIS (Infections and infestations) | 1 | 1 | 1
BRONCHITIS (Infections and infestations) | 0 | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 1
CYST (General disorders) | 2 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 7 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 2 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 6 | 0 | 0
FATIGUE (General disorders) | 5 | 0 | 0
HEADACHE (Nervous system disorders) | 6 | 0 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
MIGRAINE (Nervous system disorders) | 0 | 0 | 1
SCIATICA (Nervous system disorders) | 0 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 1
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 0 | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.